CLINICAL TRIAL: NCT07330362
Title: The Clinical Application of Artificial Intelligence Assisted Renal Biopsy Image Diagnosis System.
Brief Title: The Clinical Application of Artificial Intelligence Assisted Renal Biopsy Diagnosis System.
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024BA0045_GC
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Chronic Glomerulonephritis; Chronic Kidney Disease
Keywords: Artificial intelligence; TEM-AID; glomerulonephritis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Glomerulonephritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research project aims to collect images from patients with chronic glomerulonephritis. For each subject, the images obtained from renal biopsy will undergo evaluation by both the diagnostic model and the 'gold standard' diagnosis by pathologists. The researchers will test the subjects using the diagnostic model and compare the results with the known 'gold standard' diagnosis, in order to evaluate the AUC, specificity, and sensitivity of the diagnostic model.

DETAILED DESCRIPTION:
Renal biopsy pathology is an essential gold standard for the diagnosis of most glomerular diseases, relying on the comprehensive evaluation of H&E staining, special stains (such as PAS, PASM, and Masson), immunofluorescence, and the ultrastructural study under transmission electron microscopy (TEM). This research project aims to collect images from patients with chronic glomerulonephritis. For each subject, the images obtained from renal biopsy will undergo evaluation by both the diagnostic model and the 'gold standard' diagnosis by pathologists. The researchers will test the subjects using the diagnostic model and compare the results with the known 'gold standard' diagnosis, in order to evaluate the AUC, specificity, and sensitivity of the diagnostic model.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of informed consent form;
2. Patients clinically diagnosed or suspected of having chronic kidney disease according to the 2023 KDIGO Clinical Practice Guideline for the Evaluation and Management of Kidney Disease;
3. Undergoing renal biopsy and pathological specimen preparation.

Exclusion Criteria:

1. Biopsy tissue from donor kidney or transplanted kidney;
2. Poor quality of pathological specimen, unable to conduct pathological diagnosis.

Ages: 15 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For patients with chronic kidney disease who need further diagnosis through renal biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 2900 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The area under curve (AUC) of Receiver Operating Characteristic (ROC) curves of the TEM-AID artificial intelligence model | baseline
  The area under curve (AUC) of Receiver Operating Characteristic (ROC) curves of the TEM-AID artificial intelligence model for candidates will be calculated.

SECONDARY OUTCOMES:
The specificity of the TEM-AID artificial intelligence model. | baseline
  The specificity of the TEM-AID artificial intelligence model for candidates will be calculated.
The sensitivity of the TEM-AID artificial intelligence model. | baseline
  The sensitivity of the TEM-AID artificial intelligence model for candidates will be calculated.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanfang Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No